CLINICAL TRIAL: NCT02159053
Title: A Randomized, Double-blind, Placebo-controlled, Phase III Multicenter Study of Subcutaneous Secukinumab (150 mg) With and Without a Subcutaneous Loading Regimen to Assess Efficacy, Safety, and Tolerability up to 2 Years in Patients With Active Ankylosing Spondylitis
Brief Title: 16-week Efficacy and 2-year Safety, Tolerability and Efficacy of Secukinumab in Participants With Active Ankylosing Spondylitis
Acronym: MEASURE4
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAIN457F2320; 2013-005575-41 (EudraCT Number)
Record Dates: First submitted 2014-02-28; First posted 2014-06-09 (Estimated); Results first posted 2019-04-10 (Actual); Last update posted 2019-04-10 (Actual); Status verified 2018-11

CONDITIONS: Spondylitis, Ankylosing
Keywords: AIN457, ankylosing spondylitis, chronic inflammatory disease, inflammatory back pain, secukinumab, self-injection
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — secukinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Secukinumab 150 mg s.c. with loading (Experimental): Secukinumab 150 mg at Baseline, Weeks 1, 2, and 3, followed by dosing every four weeks starting at Week 4.
  Interventions: Biological: Secukinumab
- Secukinumab 150 mg s.c. without loading (Experimental): Secukinumab 150 mg at Baseline, followed by dosing every four weeks starting at Week 4, with Placebo at Weeks 1, 2, and 3.
  Interventions: Biological: Secukinumab
- Placebo (Placebo Comparator): Placebo at Baseline, Weeks 1, 2, 3, 4, 8, and 12, followed by dosing with Secukinumab 150 mg every four weeks starting at Week 16.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Secukinumab — Eligible subjects are randomized to each of the three treatment arms in a 1:1:1 ratio
  Other Names: Secukinumab (AIN457) 150 mg s.c.
  Arms: Secukinumab 150 mg s.c. with loading
Biological: Secukinumab — Eligible subjects are randomized to each of the three treatment arms in 1:1:1 ratio
  Other Names: Secukinumab (AIN457) 150 mg s.c.
  Arms: Secukinumab 150 mg s.c. without loading
Biological: Placebo — Eligible subjects are randomized to each of the three treatment arms in a 1:1:1 ratio
  Arms: Placebo

SUMMARY:
The purpose of this study is to provide 16-week efficacy, safety and tolerability data versus placebo to support the use of secukinumab 150 mg by subcutaneous (s.c.) self-administration with or without a loading regimen and maintenance dosing using pre-filled syringe (PFS) and to assess efficacy, safety and tolerability up to 2 years in subjects with active AS despite current or previous NSAID, non-biologic DMARD, or biologic anti-TNFα therapy.

ELIGIBILITY:
Inclusion criteria: moderate to severe AS, prior radiographic evidence according to the Modified NY Criteria (1984), inadequate response to NSAIDs.

Exclusion criteria: pregnancy or lactation, on-going infectious or malignant process on a chest X-ray or MRI, previous exposure to IL-17 or IL-17R targeting therapies, previous exposure to any biological immunomodulating agent excluding TNF antagonists, previous cell depleting therapy.

Other protocol-defined inclusion/exclusion criteria do apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2015-05-18 (Actual); Primary Completion 2016-02-23 (Actual); Study Completion 2018-01-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (80):
- United States (12):
  - Novartis Investigative Site, Anniston, Alabama
  - Novartis Investigative Site, Upland, California
  - Novartis Investigative Site, Aventura, Florida
  - Novartis Investigative Site, Peoria, Illinois
  - Novartis Investigative Site, Shreveport, Louisiana
  - Novartis Investigative Site, Lincoln, Nebraska
  - Novartis Investigative Site, Voorhees Township, New Jersey
  - Novartis Investigative Site, Oklahoma City, Oklahoma
  - Novartis Investigative Site, Duncansville, Pennsylvania
  - Novartis Investigative Site, Columbia, South Carolina
  - Novartis Investigative Site, Mesquite, Texas
  - Novartis Investigative Site, Seattle, Washington
- Australia (4):
  - Novartis Investigative Site, Kogarah, New South Wales
  - Novartis Investigative Site, Maroochydore, Queensland
  - Novartis Investigative Site, Hobart, Tasmania
  - Novartis Investigative Site, Malvern East, Victoria
- Austria (2):
  - Novartis Investigative Site, Graz
  - Novartis Investigative Site, Vienna
- Bulgaria (4):
  - Novartis Investigative Site, Pleven
  - Novartis Investigative Site, Plovdiv
  - Novartis Investigative Site, Sofia
  - Novartis Investigative Site, Targovishte
- Canada (3):
  - Novartis Investigative Site, Winnipeg, Manitoba
  - Novartis Investigative Site, Pointe-Claire, Quebec
  - Novartis Investigative Site, Trois-Rivières, Quebec
- Czechia (3):
  - Novartis Investigative Site, Ostrava, Czech Republic
  - Novartis Investigative Site, Prague, Czech Republic
  - Novartis Investigative Site, Uherské Hradiště, Czech Republic
- Denmark (2):
  - Novartis Investigative Site, Frederiksberg
  - Novartis Investigative Site, Odense
- Finland (2):
  - Novartis Investigative Site, Hyvinkää
  - Novartis Investigative Site, Jyväskylä
- Germany (12):
  - Novartis Investigative Site, Göttingen, Lower Saxony
  - Novartis Investigative Site, Bad Doberan
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Chemnitz
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Germering
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Herne
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Magdeburg
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Würzburg
- Greece (2):
  - Novartis Investigative Site, Athens
  - Novartis Investigative Site, Pátrai
- Italy (4):
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Torino, TO
  - Novartis Investigative Site, Verona, VR
- Netherlands (4):
  - Novartis Investigative Site, Amsterdam
  - Novartis Investigative Site, Heerlen
  - Novartis Investigative Site, Leiden
  - Novartis Investigative Site, Rotterdam
- Novartis Investigative Site, Kongsvinger, Norway
- Poland (4):
  - Novartis Investigative Site, Bialystok
  - Novartis Investigative Site, Elblag
  - Novartis Investigative Site, Poznan
  - Novartis Investigative Site, Warsaw
- Russia (4):
  - Novartis Investigative Site, Barnaul
  - Novartis Investigative Site, Kemerovo
  - Novartis Investigative Site, S.-Petersburg
  - Novartis Investigative Site, Saint Petersburg
- Slovakia (5):
  - Novartis Investigative Site, Piešťany, SVK
  - Novartis Investigative Site, Partizánske
  - Novartis Investigative Site, Sabinov
  - Novartis Investigative Site, Stará Ľubovňa
  - Novartis Investigative Site, Topoľčany
- Spain (7):
  - Novartis Investigative Site, Córdoba, Andalusia
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Barcelona
  - Novartis Investigative Site, Santander, Cantabria
  - Novartis Investigative Site, A Coruña, Galicia
  - Novartis Investigative Site, Santiago de Compostela, Galicia
  - Novartis Investigative Site, Barakaldo, Vizcaya
  - Novartis Investigative Site, Madrid
- Switzerland (2):
  - Novartis Investigative Site, Fribourg
  - Novartis Investigative Site, Sankt Gallen
- United Kingdom (3):
  - Novartis Investigative Site, Leytonstone, London
  - Novartis Investigative Site, Doncaster
  - Novartis Investigative Site, Wolverhampton

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Merola JF, McInnes IB, Deodhar AA, Dey AK, Adamstein NH, Quebe-Fehling E, Aassi M, Peine M, Mehta NN. Effect of Secukinumab on Traditional Cardiovascular Risk Factors and Inflammatory Biomarkers: Post Hoc Analyses of Pooled Data Across Three Indications. Rheumatol Ther. 2022 Jun;9(3):935-955. doi: 10.1007/s40744-022-00434-z. Epub 2022 Mar 19. PMID 35305260
- [Derived] Dougados M, Kiltz U, Kivitz A, Pavelka K, Rohrer S, McCreddin S, Quebe-Fehling E, Porter B, Talloczy Z. Nonsteroidal anti-inflammatory drug-sparing effect of secukinumab in patients with radiographic axial spondyloarthritis: 4-year results from the MEASURE 2, 3 and 4 phase III trials. Rheumatol Int. 2022 Feb;42(2):205-213. doi: 10.1007/s00296-021-05044-6. Epub 2021 Nov 13. PMID 34773130
- [Derived] van der Horst-Bruinsma I, Miceli-Richard C, Braun J, Marzo-Ortega H, Pavelka K, Kivitz AJ, Deodhar A, Bao W, Porter B, Pournara E. A Pooled Analysis Reporting the Efficacy and Safety of Secukinumab in Male and Female Patients with Ankylosing Spondylitis. Rheumatol Ther. 2021 Dec;8(4):1775-1787. doi: 10.1007/s40744-021-00380-2. Epub 2021 Oct 7. PMID 34618347
- [Derived] Schett G, Baraliakos X, Van den Bosch F, Deodhar A, Ostergaard M, Gupta AD, Mpofu S, Fox T, Winseck A, Porter B, Shete A, Gensler LS. Secukinumab Efficacy on Enthesitis in Patients With Ankylosing Spondylitis: Pooled Analysis of Four Pivotal Phase III Studies. J Rheumatol. 2021 Aug;48(8):1251-1258. doi: 10.3899/jrheum.201111. Epub 2021 Mar 15. PMID 33722947
- [Derived] Deodhar A, Gladman DD, McInnes IB, Spindeldreher S, Martin R, Pricop L, Porter B, Safi J Jr, Shete A, Bruin G. Secukinumab Immunogenicity over 52 Weeks in Patients with Psoriatic Arthritis and Ankylosing Spondylitis. J Rheumatol. 2020 Apr;47(4):539-547. doi: 10.3899/jrheum.190116. Epub 2019 Jun 15. PMID 31203228
- [Derived] Kivitz AJ, Wagner U, Dokoupilova E, Supronik J, Martin R, Talloczy Z, Richards HB, Porter B. Efficacy and Safety of Secukinumab 150 mg with and Without Loading Regimen in Ankylosing Spondylitis: 104-week Results from MEASURE 4 Study. Rheumatol Ther. 2018 Dec;5(2):447-462. doi: 10.1007/s40744-018-0123-5. Epub 2018 Aug 18. PMID 30121827
- See also: Introduction to clinical trials conducted by Novartis and to results of completed studies, with the aim of increasing the transparency of Novartis clinical research and making publicly available objective scientific information in a standardised format. — http://www.novartisclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 85 centers in 19 countries.
Pre-assignment Details: A total of 424 participants were screened, out of which 350 participants completed the screening phase and were randomized to three treatment groups in 1:1:1 ratio.
Groups:
- Secukinumab 150 mg With Loading Dose: Participants were subcutaneously (s.c.) administered with 150 milligrams (mg) of secukinumab at baseline, Weeks 1, 2, and 3, followed by dosing every four weeks starting at Week 4.
- Secukinumab 150 mg Without Loading Dose: Participants were s.c. administered with 150 mg of secukinumab at baseline, followed by dosing every four weeks starting at Week 4, and with Placebo at Weeks 1, 2, and 3.
- Placebo: Participants were s.c. administered with placebo matching to secukinumab at baseline, Weeks 1, 2, 3, 4, 8, and 12. Participants were further administered with 150 mg of secukinumab every four weeks starting at Week 16.
Period: Overall Study
Arm/Group | Secukinumab 150 mg With Loading Dose | Secukinumab 150 mg Without Loading Dose | Placebo
Started | 116 | 117 | 117
Paticipants Week 16 Onwards | 116 | 117 | 113
Completed | 96 | 96 | 97
Not Completed | 20 | 21 | 20
Not completed — Death | 2 | 0 | 1
Not completed — Physician Decision | 0 | 1 | 1
Not completed — Lack of Efficacy | 3 | 4 | 7
Not completed — Adverse Event | 7 | 6 | 5
Not completed — Participants/guardian decision | 8 | 10 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Secukinumab 150 mg With Loading Dose | Secukinumab 150 mg Without Loading Dose | Placebo | Total
Number analyzed (Participants) | 116 | 117 | 117 | 350
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 110 | 114 | 110 | 334
  >=65 years | 6 | 3 | 7 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.5 (11.62) | 41.2 (11.07) | 43.4 (12.46) | 43.0 (11.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 34 | 41 | 110
  Male | 81 | 83 | 76 | 240
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 2 | 0 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 2
  White | 113 | 117 | 114 | 344
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Patient's global assessment of disease activity [Mean (Standard Deviation); unit: units on a scale] — The patient's global assessment of disease activity was performed using a 0-100 millimeter (mm) VAS ranging from not severe to very severe, after the question, "How active was your disease on average during the last week?"
  units on a scale | 73.5 (15.02) | 73.2 (15.99) | 73.7 (15.05) | 73.5 (15.32)
Total back pain (0-100 mm) [Mean (Standard Deviation); unit: units on a scale] — Total back pain as measured by VAS ≥ 40 mm on a scale of 0-100 mm.
  units on a scale | 74.9 (13.07) | 74.2 (14.18) | 75 (13.8) | 74.7 (13.66)
BASDAI [Mean (Standard Deviation); unit: units on a scale] — Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) consisted of a 0 through 10 scale (0 being no problem and 10 being the worst problem, captured as a continuous VAS), which was used to answer 6 questions pertaining to the 5 major symptoms of Ankylosing Spondylitis: 1. Fatigue 2. Spinal pain 3. Joint pain / swelling 4. Areas of localized tenderness (called enthesitis, or inflammation of tendons and ligaments) 5. Morning stiffness duration 6. Morning stiffness severity.
  units on a scale | 7 (1.225) | 6.95 (1.306) | 7.06 (1.271) | 7.01 (1.265)
hs C-reactive protein [Mean (Standard Deviation); unit: Milligrams per Litre (mg/L)] — High sensitivity C-reactive protein assessment was performed in order to identify the presence of inflammation, to determine its severity, and to monitor response to treatment.
  Milligrams per Litre (mg/L) | 11.78 (18.203) | 13.84 (19.795) | 11.67 (16.699) | 12.43 (18.251)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Responded for Assessment of Spondyloarthritis International Society 20 Criteria (ASAS20) at 16 Weeks
Description: ASAS 20 response is a validated composite assessment, defined as an improvement of at least 20 percent (%) and 1 unit on a scale of 10 in three main domains and no worsening of at least 20% and 1 unit on a scale of 10 in the fourth domain within a defined time frame. Four main ASAS domains include: 1. Patient's global assessment of disease activity measured on a 100 mm VAS ranging from not severe to very severe 2. Patient's assessment of back pain, measured on a 100 mm VAS ranging from no pain to unbearable pain 3. Function represented by Bath Ankylosing Spondylitis Functional Index (BASFI) average of 10 questions regarding ability to perform specific tasks as measured by a 0-10 VAS scale 4. Inflammation represented by average of duration and severity of morning stiffness for last 2 questions on BASDAI scale (0 - no problem, 10 - worst problem)
Time Frame: 16 Weeks
Population: The analysis was performed in Full analysis set (FAS) population, defined as all participants who were randomized and received study treatment. Here, "Number of participants analysed" signifies participants evaluable for ASAS20 at Week 16.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Secukinumab 150 mg With Loading Dose | Secukinumab 150 mg Without Loading Dose | Placebo
Number analyzed (Participants) | 114 | 110 | 112
percentage of participants | 60.5 [50.9 to 69.4] | 65.5 [55.7 to 74.1] | 49.1 [49.1 to 58.7]

2. Secondary Outcome: Percentage of Participants Responded for ASAS 40 Response at 16 Weeks
Description: ASAS 20 response is a validated composite assessment, defined as an improvement of at least 40% and 2 unit on a scale of 10 in three main domains and no worsening at all in the remaining domain within a defined time frame. Four main ASAS domains include:
  1. Patient's global assessment of disease activity measured on a 100 mm VAS ranging from not severe to very severe
  2. Patient's assessment of back pain, measured on a 100 mm VAS ranging from no pain to unbearable pain
  3. Function represented by Bath Ankylosing Spondylitis Functional Index (BASFI) average of 10 questions regarding ability to perform specific tasks as measured by a 0-10 VAS scale
  4. Inflammation represented by average of duration and severity of morning stiffness for last 2 questions on BASDAI scale (0 - no problem, 10 - worst problem).
Time Frame: 16 Weeks
Population: The analysis was performed in FAS population. Here, "Number of participants analysed" signifies participants evaluable for ASAS 40 response at Week 16.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Secukinumab 150 mg With Loading Dose | Secukinumab 150 mg Without Loading Dose | Placebo
Number analyzed (Participants) | 114 | 110 | 112
percentage of participants | 39.5 [30.6 to 49.1] | 38.2 [29.2 to 48.0] | 29.5 [21.4 to 38.9]

3. Secondary Outcome: Change From Baseline in Serum High Sensitivity C-reactive Protein (hsCRP) at 16 Weeks
Description: Blood levels of C-reactive protein (CRP) is an acute phase reactant, which are indicative of inflammation and of its severity, and can be used to monitor treatment response. A hsCRP test is implemented to assess the efficacy of secukinumab (with or without load) versus placebo in reducing ankylosing spondylitis elicited systemic inflammation over the time.
Time Frame: Baseline, 16 Weeks
Population: The analysis was performed in FAS population. Here, "Number of participants analysed" signifies participants evaluable for hsCRP at Week 16.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Secukinumab 150 mg With Loading Dose | Secukinumab 150 mg Without Loading Dose | Placebo
Number analyzed (Participants) | 113 | 109 | 112
Ratio | -4.23 (15.007) | -6.57 (12.778) | 0.62 (11.699)

4. Secondary Outcome: Percentage of Participants Responded for ASAS 5/6 Response at 16 Weeks
Description: ASAS 5/6 response is a validated composite assessment, defined as an improvement of at least 20% in score in at least 5 of 6 clinical domains relevant to ankylosing spondylitis and no worsening in the remaining domain. ASAS domains includes:
  1. Patient's global assessment of disease activity measured on a 100 mm VAS ranging from not severe to very severe
  2. Patient's assessment of back pain, measured on a 100 mm VAS ranging from no pain to unbearable pain
  3. Function represented by BASFI average of 10 questions regarding ability to perform specific tasks as measured by a 0-10 VAS scale
  4. Inflammation represented by average of duration and severity of morning stiffness for last 2 questions on BASDAI scale (0 - no problem, 10 - worst problem)
  5. Spinal mobility represented by the Bath Ankylosing Spondylitis Metrology Index (BASMI) lateral spinal flexion assessment
  6. C-reactive protein (CRP, acute phase reactant).
Time Frame: 16 Weeks
Population: The analysis was performed in FAS population. Here, "Number of participants analysed" signifies participants evaluable for ASAS 5/6 response at Week 16.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Secukinumab 150 mg With Loading Dose | Secukinumab 150 mg Without Loading Dose | Placebo
Number analyzed (Participants) | 114 | 110 | 112
percentage of participants | 37.7 [29.0 to 47.3] | 45.5 [36.0 to 55.2] | 30.4 [22.2 to 39.9]

5. Secondary Outcome: Change From Baseline in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) at 16 Weeks
Description: BASDAI is a validated assessment tool using 0 through 10 scales (0 indicating "no problem" and 10 indicating "worst problem" on continuous VAS), to answer 6 questions (clinical domains) pertaining to 5 major symptoms of ankylosing spondylitis. Computed composite scores of 4 or greater indicate suboptimal disease control. BASDAI questions includes:
  1. Fatigue
  2. Spinal pain
  3. Joint pain / swelling
  4. Areas of localized tenderness (called enthesitis, or inflammation of tendons and ligaments)
  5. Morning stiffness duration
  6. Morning stiffness severity. Each symptom has equal weighting, the mean of two scores related to morning stiffness was taken (questions 5 and 6). The resulting 0 to 10 score was added to the scores from questions 1-4. The resulting 0 to 50 score was divided by 5 to give a final 0-10 BASDAI score. BASDAI was a quick and simple index taking between 30 seconds and 2 minutes for completion.
Time Frame: Baseline, 16 Weeks
Population: The analysis was performed in FAS population. Here, "Number of participants analysed" signifies participants evaluable for BASDAI at Week 16.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Secukinumab 150 mg With Loading Dose | Secukinumab 150 mg Without Loading Dose | Placebo
Number analyzed (Participants) | 114 | 110 | 112
units on a scale | -2.405 (2.1206) | -2.533 (2.1463) | -1.917 (2.2221)

6. Secondary Outcome: Change From Baseline in Physical Function Component Summary (PCS) of the Medical Outcomes Study Questionnaire Short-form Health Survey (SF-36)
Description: SF-36 is a 36 item questionnaire which measures Quality of Life across eight subscales that were scored individually: physical functioning, role- physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health. Scores are weighted sums of the questions in each section. Scores range from 0-100. Lower scores = more disability, higher scores = less disability. The overall summary scores, SF-36 physical Component Summary (PCS) was used to assess improvement from baseline in the Health-Related Quality Of Life of subjects. The change in SF-36 scores were evaluated using MMRM.
Time Frame: Baseline, 16 Weeks
Population: The analysis was performed in FAS population.Here, "Number of participants analysed" signifies participants evaluable for PCS of the SF-36 at Week 16.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Secukinumab 150 mg With Loading Dose | Secukinumab 150 mg Without Loading Dose | Placebo
Number analyzed (Participants) | 114 | 112 | 113
scores on a scale | 6.754 (6.9624) | 7.242 (8.3627) | 4.700 (7.5912)

7. Secondary Outcome: Change From Baseline in Ankylosing Spondylitis Quality of Life Questionnaire (ASQoL) at 16 Weeks
Description: ASQoL is a self-administered 18 item questionnaire that assesses disease-specific quality of life (QoL), consisting of statements that are relevant to the physical and mental conditions for a subject with ankylosing spondylitis: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each statement is answered as a 'Yes' (scored as 1) or 'No' (scored as 0). All item scores are summed to give a total score. Total score ranges from 0 (good QoL) to 18 (poor QoL). The change in ASQoL scores was evaluated using a mixed effect repeated measures model (MMRM).
Time Frame: Baseline, 16 Weeks
Population: The analysis was performed in FAS population. Here, "Number of participants analysed" signifies participants evaluable for ASQoL at Week 16.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Secukinumab 150 mg With Loading Dose | Secukinumab 150 mg Without Loading Dose | Placebo
Number analyzed (Participants) | 114 | 112 | 113
units on a scale | -4.2 (4.63) | -4.7 (5.05) | -3.0 (4.74)

8. Secondary Outcome: Number of Participants With Adverse Events (AEs), Deaths, Serious Adverse Events (SAEs) and Related Discontinuations at 104 Weeks
Description: AEs were defined as any unfavorable and unintended diagnosis, symptom, sign (including an abnormal laboratory finding), syndrome or disease which either occurs during study, having been absent at baseline, or, if present at baseline, appears to worsen. SAEs were defined as any untoward medical occurrences that result in death, are life threatening, require (or prolong) hospitalization, cause persistent or significant disability/incapacity, result in congenital anomalies or birth defects, or are other conditions which in judgement of investigators represent significant hazards.
Time Frame: 104 Weeks
Population: The analysis was performed on the safety population, defined as all participants who took at least one dose of study treatment during the treatment period.
Measure: Number; unit: participants
Groups:
- All Secukinumab 150 mg Treated Participants: All participants who were s.c. administered with secukinumab during the study.
Arm/Group | Secukinumab 150 mg With Loading Dose | Secukinumab 150 mg Without Loading Dose | Placebo | All Secukinumab 150 mg Treated Participants
Number analyzed (Participants) | 116 | 117 | 117 | 346
participants
  AEs | 100 | 98 | 65 | 289
  SAEs | 16 | 11 | 4 | 39
  Death | 2 | 0 | 0 | 4
  Discontinued study treatment due to any AEs | 9 | 5 | 1 | 20

9. Secondary Outcome: Percentage of Participants Responded for ASAS 20 at Week 4
Description: ASAS 20 response is a validated composite assessment, defined as an improvement of at least 20% and 1 unit on a scale of 10 in three main domains and no worsening of at least 20% and 1 unit on a scale of 10 in the fourth domain within a defined time frame. Four main ASAS domains include:
  1. Patient's global assessment of disease activity measured on a 100 mm VAS ranging from not severe to very severe
  2. Patient's assessment of back pain, measured on a 100 mm VAS ranging from no pain to unbearable pain
  3. Function represented by Bath Ankylosing Spondylitis Functional Index (BASFI) average of 10 questions regarding ability to perform specific tasks as measured by a 0-10 VAS scale
  4. Inflammation represented by average of duration and severity of morning stiffness for last 2 questions on BASDAI scale (0 - no problem, 10 - worst problem).
Time Frame: Week 4
Population: The analysis was performed in FAS population. Here, "Number of participants analysed" signifies participants evaluable for ASAS 20 at Week 16.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Secukinumab 150 mg With Loading Dose | Secukinumab 150 mg Without Loading Dose | Placebo
Number analyzed (Participants) | 116 | 114 | 115
percentage of participants | 49.1 [39.8 to 58.5] | 55.3 [45.7 to 64.6] | 40.0 [31.1 to 49.6]

10. Secondary Outcome: Percentage of Participants Responded for ASAS 40 Response at Week 4
Description: as for outcome 2
Time Frame: Week 4
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Secukinumab 150 mg With Loading Dose | Secukinumab 150 mg Without Loading Dose | Placebo
Number analyzed (Participants) | 116 | 114 | 115
percentage of participants | 29.3 [21.4 to 38.6] | 27.2 [19.5 to 36.5] | 18.3 [11.9 to 26.8]

ADVERSE EVENTS:
Time Frame: Adverse Events and Serious Adverse Events were collected for the maximum actual duration of treatment exposure and follow up for a participant per the protocol for approximately 104 weeks.
Description: Serious Adverse Events are monitored from date of First Participant First Visit (FPFV) until Last Participant Last Visit (LPLV). All other adverse events are monitored from First Participant First Treatment until LPLV.
Groups:
- Secukinumab 150 mg With Loading: Participants were s.c. administered with 150 mg of secukinumab at baseline, Weeks 1, 2, and 3, followed by dosing every four weeks starting at Week 4.
Arm/Group | Secukinumab 150 mg Without Loading Dose | Secukinumab 150 mg With Loading | All Secukinumab 150 mg Treated Participants | Placebo
All-Cause Mortality (participants affected / at risk) | 2/116 | 0/117 | 4/346 | 0/117
Serious Adverse Events (participants affected / at risk) | 18/116 | 11/117 | 43/346 | 4/117
Other Adverse Events (participants affected / at risk) | 90/116 | 89/117 | 254/346 | 54/117
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Secukinumab 150 mg Without Loading Dose (N=116) | Secukinumab 150 mg With Loading (N=117) | All Secukinumab 150 mg Treated Participants (N=346) | Placebo (N=117)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiac failure acute (Cardiac disorders) | 1 | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 1 | 0
Pericarditis (Cardiac disorders) | 1 | 0 | 1 | 0
Acute vestibular syndrome (Ear and labyrinth disorders) | 1 | 0 | 1 | 0
Papilloedema (Eye disorders) | 0 | 1 | 1 | 0
Retinal detachment (Eye disorders) | 0 | 1 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Anal fistula (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0 | 2 | 0
Crohn's disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Duodenitis (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Gastritis erosive (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Fatigue (General disorders) | 1 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 2 | 0
Atypical pneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Chronic tonsillitis (Infections and infestations) | 0 | 1 | 1 | 0
Erysipelas (Infections and infestations) | 2 | 0 | 3 | 0
Otitis media acute (Infections and infestations) | 1 | 0 | 1 | 0
Tinea pedis (Infections and infestations) | 0 | 0 | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Tendon injury (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 1 | 0
Weight decreased (Investigations) | 1 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Femoroacetabular impingement (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Myofascial pain syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2 | 0
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Testis cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 2 | 0
Basal ganglia haemorrhage (Nervous system disorders) | 0 | 0 | 1 | 0
Migraine (Nervous system disorders) | 0 | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 1 | 0
VIth nerve paralysis (Nervous system disorders) | 0 | 1 | 1 | 0
Depression suicidal (Psychiatric disorders) | 0 | 0 | 1 | 0
Somatic symptom disorder (Psychiatric disorders) | 0 | 1 | 1 | 0
Bladder diverticulum (Renal and urinary disorders) | 0 | 0 | 1 | 0
Glomerulonephritis membranous (Renal and urinary disorders) | 0 | 1 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1 | 1 | 0
Renal colic (Renal and urinary disorders) | 0 | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0 | 1 | 0
Rectocele (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Peripheral artery occlusion (Vascular disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Secukinumab 150 mg Without Loading Dose (N=116) | Secukinumab 150 mg With Loading (N=117) | All Secukinumab 150 mg Treated Participants (N=346) | Placebo (N=117)
Anaemia (Blood and lymphatic system disorders) | 1 | 3 | 5 | 0
Leukopenia (Blood and lymphatic system disorders) | 4 | 1 | 8 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 7 | 0
Atrioventricular block first degree (Cardiac disorders) | 4 | 1 | 8 | 0
Vertigo (Ear and labyrinth disorders) | 3 | 3 | 7 | 0
Iridocyclitis (Eye disorders) | 3 | 1 | 7 | 0
Iritis (Eye disorders) | 1 | 3 | 7 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 3 | 8 | 0
Abdominal pain upper (Gastrointestinal disorders) | 6 | 1 | 10 | 0
Diarrhoea (Gastrointestinal disorders) | 9 | 11 | 28 | 6
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 3 | 5 | 0
Mouth ulceration (Gastrointestinal disorders) | 3 | 2 | 6 | 1
Nausea (Gastrointestinal disorders) | 8 | 1 | 13 | 2
Toothache (Gastrointestinal disorders) | 2 | 3 | 5 | 0
Fatigue (General disorders) | 4 | 3 | 8 | 4
Influenza like illness (General disorders) | 2 | 3 | 5 | 0
Non-cardiac chest pain (General disorders) | 0 | 3 | 4 | 1
Pyrexia (General disorders) | 3 | 1 | 8 | 1
Bronchitis (Infections and infestations) | 13 | 8 | 31 | 1
Ear infection (Infections and infestations) | 3 | 0 | 4 | 0
Fungal skin infection (Infections and infestations) | 5 | 1 | 7 | 0
Gastroenteritis (Infections and infestations) | 5 | 3 | 10 | 2
Herpes simplex (Infections and infestations) | 3 | 1 | 5 | 0
Influenza (Infections and infestations) | 7 | 9 | 19 | 5
Laryngitis (Infections and infestations) | 3 | 2 | 7 | 0
Nasopharyngitis (Infections and infestations) | 32 | 29 | 80 | 10
Oral herpes (Infections and infestations) | 4 | 3 | 9 | 2
Pharyngitis (Infections and infestations) | 2 | 6 | 10 | 3
Pulpitis dental (Infections and infestations) | 3 | 0 | 3 | 0
Respiratory tract infection (Infections and infestations) | 6 | 10 | 22 | 3
Rhinitis (Infections and infestations) | 3 | 7 | 15 | 1
Sinusitis (Infections and infestations) | 4 | 4 | 9 | 0
Tonsillitis (Infections and infestations) | 1 | 3 | 10 | 0
Tooth infection (Infections and infestations) | 3 | 0 | 4 | 0
Upper respiratory tract infection (Infections and infestations) | 11 | 17 | 37 | 6
Urinary tract infection (Infections and infestations) | 3 | 2 | 7 | 0
Contusion (Injury, poisoning and procedural complications) | 4 | 4 | 10 | 0
Fall (Injury, poisoning and procedural complications) | 4 | 0 | 5 | 1
Alanine aminotransferase increased (Investigations) | 5 | 4 | 10 | 1
Aspartate aminotransferase increased (Investigations) | 3 | 4 | 8 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 1 | 3 | 3
Hyperlipidaemia (Metabolism and nutrition disorders) | 6 | 1 | 9 | 1
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 12 | 11 | 29 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 11 | 15 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 3 | 4 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 7 | 23 | 5
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 6 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 2 | 8 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 | 0 | 5 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 5 | 10 | 0
Spondylitis (Musculoskeletal and connective tissue disorders) | 1 | 3 | 4 | 1
Headache (Nervous system disorders) | 10 | 2 | 18 | 5
Depression (Psychiatric disorders) | 0 | 5 | 6 | 0
Haematuria (Renal and urinary disorders) | 0 | 3 | 3 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 4 | 18 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 | 5 | 16 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 5 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 4 | 6 | 2
Eczema (Skin and subcutaneous tissue disorders) | 4 | 3 | 7 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 3 | 8 | 2
Rash (Skin and subcutaneous tissue disorders) | 3 | 3 | 9 | 0
Hypertension (Vascular disorders) | 9 | 6 | 18 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.